CLINICAL TRIAL: NCT01614795
Title: A Phase II Study of Cixutumumab (IMC-A12) in Combination With Temsirolimus in Pediatric Patients With Recurrent or Refractory Solid Tumors
Brief Title: Cixutumumab and Temsirolimus in Treating Younger Patients With Recurrent or Refractory Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01971; NCI-2012-01971 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ADVL1221; COG-ADVL1221; CDR0000734871; ADVL1221 (Other: Childrens Oncology Group); ADVL1221 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Results first posted 2015-03-31 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Childhood Alveolar Soft Part Sarcoma; Childhood Angiosarcoma; Childhood Epithelioid Sarcoma; Childhood Fibrosarcoma; Childhood Gliosarcoma; Childhood Leiomyosarcoma; Childhood Liposarcoma; Childhood Malignant Peripheral Nerve Sheath Tumor; Childhood Synovial Sarcoma; Previously Treated Childhood Rhabdomyosarcoma; Recurrent Childhood Rhabdomyosarcoma; Recurrent Childhood Soft Tissue Sarcoma; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Osteosarcoma; Rhabdomyosarcoma
MeSH Terms: conditions — Hemangiosarcoma; Sarcoma; Fibrosarcoma; Liposarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Osteosarcoma; Rhabdomyosarcoma | interventions — cixutumumab; temsirolimus; Sirolimus

ARMS (1):
- Treatment (cixutumumab, temsirolimus) (Experimental): Patients receive cixutumumab IV over 1 hour and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 25 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cixutumumab; Other: Laboratory Biomarker Analysis; Drug: Temsirolimus

INTERVENTIONS:
Biological: Cixutumumab — Given IV
  Other Names: Anti-IGF-1R Recombinant Monoclonal Antibody IMC-A12; IMC-A12
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel

SUMMARY:
This phase II trial studies how well cixutumumab and temsirolimus work in treating patients with recurrent or refractory sarcoma. Monoclonal antibodies, such as cixutumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving cixutumumab and temsirolimus together may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate to the combination of cixutumumab and temsirolimus in patients with relapsed or refractory osteosarcoma, Ewing sarcoma, rhabdomyosarcoma, or non-rhabdomyosarcoma soft tissue sarcoma.

II. To further describe the toxicities (including dose-limiting toxicities) of cixutumumab and temsirolimus administered on this schedule.

SECONDARY OBJECTIVES:

I. To assess the progression-free survival for patients treated in each disease stratum with this drug combination.

II. To assess the incidence of insulin-like growth factor 1 receptor (IGF-1R), insulin receptor, ERK, RON, and mammalian target of rapamycin (mTOR) pathway activation in archival tumor material, and correlate with response.

III. To evaluate minimal residual disease and IGF-1R tumor cell expression in the blood and bone marrow of Ewing sarcoma patients using flow cytometry.

OUTLINE: This is a multicenter study. Patients are stratified according to diagnosis (osteosarcoma vs Ewing sarcoma/PNET vs rhabdomyosarcoma vs non-rhabdomyosarcoma soft tissue sarcoma).

Patients receive cixutumumab IV over 1 hour and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 25 courses in the absence of disease progression or unacceptable toxicity.

Archived tumor tissue samples from most recent biopsy are collected and analyzed for IGF-1R, insulin receptor, AKT, ERK, mTOR, and S6 kinase pathway activation by immunohistochemistry (IHC) and banked for future correlative studies. Blood and bone marrow samples, from patients with Ewing sarcoma, may be collected at baseline and periodically during treatment for minimal residual disease analysis by flow cytometry.

After completion of study treatment, patients are followed up periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any of the following tumors who have experienced relapse following front-line therapy, or who are refractory to front-line therapy, are eligible:

  * Osteosarcoma
  * Ewing sarcoma/peripheral primitive neuroectodermal tumor (PNET)
  * Rhabdomyosarcoma
  * Non-rhabdomyosarcoma soft tissue sarcoma
* Patients must have had histologic verification of malignancy at original diagnosis or relapse
* All patients are required to submit archival tumor samples for immunohistochemical analysis (either paraffin-embedded tumor blocks or unstained slides)

  * Tissue samples collected at original diagnosis or at relapse or at any subsequent resections or biopsies should be available and ready for shipment to the Biopathology Center (BPC) at time of study enrollment; the samples are required even if tissue samples have previously been sent to the BPC for other purposes or studies; blocks or slides should be shipped to the BPC within 7 days of study enrollment
* Patients must have radiographically measurable disease

  * Measurable disease is defined as the presence of at least one lesion on magnetic resonance imaging (MRI) or computed tomography (CT) scan that can be accurately measured with the longest diameter a minimum of 10 mm in at least one dimension (CT scan slice thickness no greater than 5 mm)
  * The following do not qualify as measurable disease:

    * Malignant fluid collections (e.g., ascites, pleural effusions)
    * Bone marrow infiltration
    * Lesions only detected by nuclear medicine studies (e.g., bone, gallium, or positron emission tomography [PET] scans)
    * Elevated tumor markers in plasma or cerebrospinal fluid(CSF)
    * Previously radiated lesions that have not demonstrated clear progression post radiation
    * Leptomeningeal lesions that do not meet the measurements noted above
* Patient?s current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Patients with known central nervous system metastases are excluded unless treated surgically or with radiotherapy and stable with no recurrent lesions for at least 3 months
* Patients must have a Lansky or Karnofsky performance status score of ? 50%, corresponding to Eastern Cooperative Oncology Group (ECOG) categories 0, 1, or 2; use Karnofsky for patients > 16 years of age and Lansky for patients ? 16 years of age

  * Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* For patients with solid tumors without bone marrow involvement:

  * Peripheral absolute neutrophil count (ANC) ? 1,000/?L
  * Platelet count ? 100,000/?L (transfusion independent, defined as not receiving platelet transfusions within a 7-day period prior to enrollment)
  * Hemoglobin ? 8.0 g/dL (may receive red blood cell [RBC] transfusions)
* For patients with solid tumors and known bone marrow metastatic disease:

  * ANC ? 750/?L
  * Platelet count ? 50,000/?L (may receive platelet transfusions)
  * Hemoglobin ? 8.0 g/dL (may receive RBC transfusions)

    * For patients with known bone marrow metastatic disease, transfusions are permitted to meet both platelet and hemoglobin criteria; patients must not be known to be refractory to red blood cell or platelet transfusions
* Creatinine clearance or radioisotope GFR ? 70 mL/min OR a serum creatinine based on age/gender as follows:

  * 0.6 mg/dL (1 to < 2 years of age)
  * 0.8 mg/dL (2 to < 6 years of age)
  * 1.0 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (males) or 1.4 mg/dL (females) (13 to < 16 years of age)
  * 1.7 mg/dL (males) or 1.4 mg/dL (females) ( ? 16 years of age)
* Total bilirubin ? 1.5 times upper limit of normal (ULN)
* Serum glutamic pyruvate transaminase(SGPT) (alanine aminotransaminase [ALT]) ? 2.5 times ULN (for the purpose of this study, the ULN for SGPT is 45 U/L)
* Serum albumin ? 2 g/dL
* Patients with seizure disorder may be enrolled if receiving non-enzyme-inducing anticonvulsants and well controlled
* Patients with known type I or type II diabetes mellitus are not eligible
* Serum glucose values must be within the normal limits for age; if the initial blood glucose is a random sample that is outside normal limits, then a follow-up fasting blood glucose should be obtained and must be within the normal limits for age
* Serum cholesterol levels must be < grade 2 (< 300 mg/dL), and serum triglyceride levels must be < grade 2 (< 2.5 times ULN)
* Patients who are pregnant or breast-feeding are not eligible for this study
* Negative pregnancy tests must be obtained in girls who are post-menarchal
* Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for the duration of the study and for 3 months after the last dose of cixutumumab
* Patients who have an uncontrolled infection are not eligible
* Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study are not eligible
* See Disease Characteristics
* There is no limit to the number of prior treatment regimens; however, patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to study enrollment
* Patients must not have received myelosuppressive chemotherapy within 3 weeks of enrollment (6 weeks if prior nitrosourea)
* At least 7 days must have elapsed since the completion of therapy with a growth factor; at least 14 days must have elapsed after receiving pegfilgrastim
* At least 7 days must have elapsed since the completion of therapy with a biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period prior to enrollment must be extended beyond the time during which adverse events are known to occur
* At least 3 half-lives must have elapsed since prior therapy that included a monoclonal antibody
* ? 2 weeks must have elapsed since local palliative radiotherapy (XRT) (small port); 3 months must have elapsed if 50% radiation of pelvis; 6 weeks must have elapsed if therapeutic doses of metaiodobenzylguanidine(MIBG) or other substantial bone marrow irradiation was given
* No evidence of active graft-vs-host disease and 2 months must have elapsed since stem cell transplant or rescue
* Growth factors that support platelet or white cell number or function must not have been administered within the 7 days prior to enrollment (14 days if Neulasta?)
* Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for the 7 days prior to enrollment are not eligible
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents, including chemotherapy, radiotherapy, immunotherapy, or biologic therapy, are not eligible
* Patients receiving insulin or growth hormone therapy are not eligible
* Patients who are receiving enzyme-inducing anticonvulsants are not eligible
* Use of warfarin is not allowed while on study; patients already on warfarin should use alternative anticoagulants while on this study; warfarin must not have been administered within 7 days of starting protocol therapy
* Patients who have received prior therapy targeting IGF-1R with either monoclonal antibodies or small molecule tyrosine kinase inhibitors are NOT eligible
* Prior treatment with mTOR inhibitors (e.g., rapamycin, temsirolimus, everolimus, deforolimus) is NOT allowed
* Patients who have had major surgery within 3 weeks prior to enrollment are not eligible; procedures such as placement of a central vascular catheter or limited tumor biopsy are not considered major surgery

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2012-06-18 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2014-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Wagner, Principal Investigator — Children's Oncology Group
Locations (76):
- United States (74):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Palmetto Health Richland, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Marshfield Clinic, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The analysis strategy for secondary outcome measures accommodates the possibility that the Progression-Free Interval and IHC could have different statistical characteristics across the different histologies that define the study groups.
Groups:
- Group 1 Relapsed or Refractory Osteosarcoma; Group 2 Relapsed or Refractory Ewing Sarcoma/Peripheral PNET; Group 3 Relapsed or Refractory Rhabdomyosarcoma; Group 4 Relapsed or Refractory Non-rhabdo Soft Tissue Sarcoma: Patients receive cixutumumab IV over 1 hour and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 25 courses in the absence of disease progression or unacceptable toxicity.
  cixutumumab: Given IV, Days 1, 8, 15, and 22, dosage 6 mg/kg. Cixutumumab dose is based on weight (kg).
  temsirolimus: Given IV, Days 1, 8, 15, and 22 8 mg/m2 (maximum dose = 16 mg) (Cycle 1), Dose escalation to 10 mg/m2 (maximum dose = 20 mg). Temsirolimus dose is based on BSA.
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Group 1 Relapsed or Refractory Osteosarcoma | Group 2 Relapsed or Refractory Ewing Sarcoma/Peripheral PNET | Group 3 Relapsed or Refractory Rhabdomyosarcoma | Group 4 Relapsed or Refractory Non-rhabdo Soft Tissue Sarcoma
Started | 11 | 12 | 11 | 12
Completed | 0 | 0 | 0 | 0
Not Completed | 11 | 12 | 11 | 12
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 10 | 10 | 9 | 8
Not completed — Physician Decision | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2
Not completed — Ineligible | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 Relapsed or Refractory Osteosarcoma | Group 2 Relapsed or Refractory Ewing Sarcoma/Peripheral PNET | Group 3 Relapsed or Refractory Rhabdomyosarcoma | Group 4 Relapsed or Refractory Non-rhabdo Soft Tissue Sarcoma | Total
Number analyzed (Participants) | 11 | 12 | 11 | 12 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 8 | 9 | 7 | 31
  Between 18 and 65 years | 4 | 4 | 2 | 5 | 15
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 18 [7 to 25] | 17.5 [9 to 27] | 14 [1 to 23] | 17.5 [13 to 26] | 17 [1 to 27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 8 | 5 | 20
  Male | 10 | 6 | 3 | 7 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 3 | 0 | 4
  Not Hispanic or Latino | 10 | 12 | 8 | 11 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 0 | 2
  Black or African American | 2 | 0 | 0 | 1 | 3
  White | 7 | 8 | 9 | 7 | 31
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 11 | 12 | 45
  Canada | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (PR or CR) by Response Evaluation Criteria in Solid Tumors (RECIST).
Description: Per Response evaluation criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions. Overall Response (OR)= CR+PR. The combination of sufficient activity is considered if the true response rate is 35% or greater.
Time Frame: 6 cycles (168 days)
Population: One (1) of the patients in Group 1 and one (1) of the patients in Group 4 were considered inevaluable for response assessment. One (1) of the patients in Group 2 was ineligible.
Measure: Number; unit: participants
Arm/Group | Group 1 Relapsed or Refractory Osteosarcoma | Group 2 Relapsed or Refractory Ewing Sarcoma/Peripheral PNET | Group 3 Relapsed or Refractory Rhabdomyosarcoma | Group 4 Relapsed or Refractory Non-rhabdo Soft Tissue Sarcoma
Number analyzed (Participants) | 10 | 11 | 11 | 11
participants
  Non-Responder | 10 | 11 | 11 | 11
  Responder | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Cycles of Toxicity
Description: The number of patients-cycles where CTC Version 4 grade 3 or higher increased Alanine aminotransferase was observed
Time Frame: Duration of protocol therapy - Up to 25 cycles (700 days)
Population: One hundred six (106) cycles were reported for the analysis of this toxicity
Measure: Number; unit: cycles
Units Other Than Participants: cycles
Arm/Group | Treatment (Cixutumumab, Temsirolimus)
Number analyzed (Participants) | 46
Number analyzed (cycles) | 106
cycles
  Alkaline phosphatase | 1
  Anaphylaxis | 1
  Anemia | 3
  Ascites | 1
  Aspartate aminotransferase | 3
  Decreased lymphocyte count | 1
  Decreased platelet count | 5
  Decreased white blood cells | 3
  Duodenal obstruction | 1
  Epistaxis | 1
  Extremity pain | 1
  Hyperglycemia | 1
  Hypermagnesemia | 1
  Hypertriglyceridemia | 2
  Hyperuricemia | 1
  Hypoalbuminemia | 1
  Hypokalemia | 5
  Hyponatremia | 1
  Hypophosphatemia | 4
  Hypoxia | 1
  Increased alanine aminotransferase | 2
  Increased blood bilirubin | 1
  Increased creatinine | 1
  Multi-organ failure | 1
  Neutopenia | 6
  Non-cardiac chest pain | 1
  Other cardiac disorders | 1
  Other infections and infestations | 1
  Oral mucocitis | 4
  Pain | 2
  Paronychia | 1
  Urinary tract infection | 1
  Urinary tract obstruction | 1
  Weight loss | 1
  Wound infection | 1

3. Secondary Outcome: Progression-free Interval
Description: Percentage Probability of remaining progression-free 5 years after enrollment estimated by the method of Kaplan and Meier
Time Frame: 10 months after enrollment
Population: The 10 month time point was chosen since the shortest follow-up available was observed in Group 3 (relapsed or refractory rhabdomyosarcoma) where the last patient under observation was censored after completing 10 months of follow-up
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Group 1 Relapsed or Refractory Osteosarcoma | Group 2 Relapsed or Refractory Ewing Sarcoma/Peripheral PNET | Group 3 Relapsed or Refractory Rhabdomyosarcoma | Group 4 Relapsed or Refractory Non-rhabdo Soft Tissue Sarcoma
Number analyzed (Participants) | 10 | 11 | 11 | 11
percent probability | 9.09 [0.54 to 33.29] | 9.09 [0.54 to 33.29] | 9.09 [0.54 to 33.29] | 16.67 [2.65 to 41.30]

4. Secondary Outcome: Expression Levels of IGF-1R, Insulin Receptor, ERK, RON, and mTOR
Description: Number of patients expressing insulin-like growth factor 1 receptor (IGF-1R), insulin receptor, ERK, RON, and mammalian target of rapamycin (mTOR) at levels 0, 1+, 2+, 3+ by immunohistochemistry.
Time Frame: Baseline
Population: All specimens for the IHC analysis for IGF-1R, Insulin Receptor, ERK, RON, and mTOR were obtained prior to the start of treatment on ADVL1221. Levels 0, 1+, 2+ and 3+ represent increasing strengths of IHC staining.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Relapsed or Refractory Osteosarcoma | Group 2 Relapsed or Refractory Ewing Sarcoma/Peripheral PNET | Group 3 Relapsed or Refractory Rhabdomyosarcoma | Group 4 Relapsed or Refractory Non-rhabdo Soft Tissue Sarcoma
Number analyzed (Participants) | 10 | 11 | 11 | 11
Participants
  IGF-1R level 0 | 2 | 4 | 1 | 3
  IGF-1R level 1+ | 4 | 3 | 0 | 4
  IGF-1R level 2+ | 2 | 2 | 2 | 5
  IGF-1R level 3+ | 2 | 2 | 8 | 1
  Insulin receptor level 0: number analyzed (Participants) | 9 | 11 | 11 | 11
  Insulin receptor level 0 | 4 | 4 | 4 | 3
  Insulin receptor level 1+: number analyzed (Participants) | 9 | 11 | 11 | 11
  Insulin receptor level 1+ | 2 | 2 | 1 | 2
  Insulin receptor level 2+: number analyzed (Participants) | 9 | 11 | 11 | 11
  Insulin receptor level 2+ | 2 | 3 | 4 | 2
  Insulin receptor level 3+: number analyzed (Participants) | 9 | 11 | 11 | 11
  Insulin receptor level 3+ | 1 | 2 | 2 | 2
  ERK level 0 | 2 | 5 | 6 | 3
  ERK level 1+ | 5 | 5 | 2 | 4
  ERK level 2+ | 1 | 0 | 3 | 3
  ERK Level 3+ | 2 | 1 | 0 | 1
  RON level 0 | 7 | 10 | 10 | 6
  RON level 1+ | 3 | 1 | 1 | 4
  RON level 2+ | 0 | 0 | 0 | 0
  RON level 3+ | 0 | 0 | 0 | 1
  mTOR level 0 | 8 | 7 | 10 | 8
  mTOR level 1+ | 2 | 3 | 1 | 3
  mTOR level 2+ | 0 | 1 | 0 | 0
  mTOR level 3+ | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Patients With Detectable Bone Marrow Micrometastatic Disease Estimated as the Proportion of Eligible Patients Entered Into the Ewing Sarcoma Stratum Who Have Detectable Tumor Cells in the Marrow at Enrollment
Time Frame: Baseline
Population: 2 patients of the 12 patients enrolled in the Ewing Sarcoma stratum submitted specimens for analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cixutumumab, Temsirolimus)
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Description: SAE field contains NCI Common Toxicity Criteria for Adverse Events (CTCAEs) submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs.
Arm/Group | Group 1 Relapsed or Refractory Osteosarcoma | Group 2 Relapsed or Refractory Ewing Sarcoma/Peripheral PNET | Group 3 Relapsed or Refractory Rhabdomyosarcoma | Group 4 Relapsed or Refractory Non-rhabdo Soft Tissue Sarcoma
Serious Adverse Events (participants affected / at risk) | 2/11 | 3/11 | 2/11 | 7/12
Other Adverse Events (participants affected / at risk) | 11/11 | 5/11 | 7/11 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 Relapsed or Refractory Osteosarcoma (N=11) | Group 2 Relapsed or Refractory Ewing Sarcoma/Peripheral PNET (N=11) | Group 3 Relapsed or Refractory Rhabdomyosarcoma (N=11) | Group 4 Relapsed or Refractory Non-rhabdo Soft Tissue Sarcoma (N=12)
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 0
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Anaphylaxis (Immune system disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0
Cardiac disorders - Other (Cardiac disorders) | 0 | 0 | 0 | 1
Creatinine increased (Investigations) | 0 | 0 | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fever (General disorders) | 0 | 0 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Infections and infestations - Other (Infections and infestations) | 0 | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Multi-organ failure (General disorders) | 0 | 0 | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Weight loss (Investigations) | 1 | 0 | 0 | 0
White blood cell decreased (Investigations) | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 Relapsed or Refractory Osteosarcoma (N=11) | Group 2 Relapsed or Refractory Ewing Sarcoma/Peripheral PNET (N=11) | Group 3 Relapsed or Refractory Rhabdomyosarcoma (N=11) | Group 4 Relapsed or Refractory Non-rhabdo Soft Tissue Sarcoma (N=12)
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0
Creatinine increased (Investigations) | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 5 | 1 | 3 | 3
Neutrophil count decreased (Investigations) | 3 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 2 | 3 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
White blood cell decreased (Investigations) | 2 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less